CLINICAL TRIAL: NCT05114018
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Effects of 'Next Generation Beneficial Microbes', Akkermansia Muciniphila (AMF-01), on Long-term Improvements in Insulin Resistance in Otherwise Healthy Hyperglycaemic Adults
Brief Title: Effect of Pasteurized Akkermansia Muciniphila on Insulin Resistance in Otherwise Healthy Subjects With Dysglycaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A-Mansia Biotech S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFCRO-117
Record Dates: First submitted 2021-10-07; First posted 2021-11-09 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2023-09

CONDITIONS: Metabolic Syndrome; Pre-diabetes; Overweight and Obesity
MeSH Terms: conditions — Metabolic Syndrome; Glucose Intolerance; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel group, multi-center trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group receiving pasteurized Akkermansia muciniphila (Experimental): Experimental group receiving pasteurized Akkermansia muciniphila.
  Interventions: Dietary Supplement: Pasteurized A. muciniphila
- Control group (Placebo Comparator): Control group receiving placebo, identical to verum regarding the form, size, taste, color and intake.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Pasteurized A. muciniphila — Daily oral dose
  Arms: Experimental group receiving pasteurized Akkermansia muciniphila
Dietary Supplement: placebo — Placebo = identical to verum regarding the form, size, taste, color and intake
  Arms: Control group

SUMMARY:
The purpose of this study is to demonstrate the efficacy of pasteurized Akkermansia muciniphila (pAKK) in improving insulin sensitivity in hyperglycaemic, but otherwise healthy persons with metabolic syndrome. This is the primary objective of this study. Secondary objectives consist of evaluation of the effects of next generation beneficial microbes on metabolic health, anthropometry and body composition, and safety.

Therefore, the trial is designed as a phase 2, randomized, double-blind, placebo-controlled, parallel group, multi-center trial comparing pAKK with placebo in restoring insulin sensitivity in dysglycaemic but otherwise healthy subjects with metabolic syndrome.

In total, 144 enrolled participants will attend 6 study visits in total. Study visits may be conducted in the clinic, at home by a Healthcare Professional, or by telephone / telemedicine.

DETAILED DESCRIPTION:
Overweight and obesity have reached worldwide epidemic level. Observation of elevated glycaemia like impaired fasting glucose and impaired glucose tolerance are reflecting pre-diabetic states often occurring in the context of development of insulin resistance in persons with metabolic syndrome. Moreover, this status is associated with the risk for developing type 2 diabetes as well as cardiovascular disease. In a proof of concept study the supplementation with A. muciniphila was safe and improved metabolic health in persons with metabolic syndrome.

The purpose of this study is to demonstrate the efficacy of pasteurized Akkermansia muciniphila (pAKK) in improving insulin sensitivity in hyperglycaemic, but otherwise healthy persons with metabolic syndrome. This is the primary objective of this study. Secondary objectives consist of evaluation of the effects of next generation beneficial microbes on metabolic health, anthropometry and body composition, and safety.

Therefore, the trial is designed as a phase 2, randomized, double-blind, placebo-controlled, parallel group, multi-center trial comparing pAKK with placebo in restoring insulin sensitivity in dysglycaemic but otherwise healthy subjects with metabolic syndrome.

In total, 144 enrolled participants will attend 6 study visits in total. Study visits may be conducted in the clinic, at home by a Healthcare Professional, or by telephone / telemedicine.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent;
* BMI between >25 and <40 Kg/m2;
* Qualifying for the diagnosis of metabolic syndrome according to the International Diabetes Federation (IDF 2006) criteria. At least any three of five citeria, with the modification that the criterion FPG≥100 mg/dL (5.6 mmol/L) is required among at least three of five:

  * Increased waist circumference: for Europid, sub-Saharan African, Eastern and Middle-Eastern ≥94 cm (men) or ≥80 cm (women), with ethnic-specific waist circumference cut-points: for South Asian and Chinese patients, waist ≥90 cm (men) or ≥80 cm (women); for Japanese patients, waist ≥90 cm (men) or ≥80 cm (women);
  * Triglycerides ≥150 mg/dL (1.7 mmol/L) (exception: triglycerides ≥100 mg/dL (1.13mmol/L) for sub-Saharan African) or treatment for elevated triglycerides;
  * HDL cholesterol <40 mg/dL (1.03 mmol/L) in men or <50 mg/dL (1.29 mmol/L) in females, or treatment for low HDL;
  * Systolic blood pressure ≥130, diastolic blood pressure ≥85 mmHg, or treatment for hypertension;
  * FPG ≥100 mg/dL (5.6 mmol/L) or previously diagnosed type 2 diabetes; an oral glucose tolerance test is recommended for patients with an elevated FPG, but it is not required.
* If participant has a prior diagnosis of pre-diabetes or Type II diabetes, and has been unmedicated for 3-months prior to screening;
* If female, must meet all the following criteria:

  * Not pregnant or breastfeeding
  * If of childbearing potential (including peri-menopausal women who have had a menstrual period within one year) must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as double barrier methods [male condom with spermicide, with or without cervical cap or diaphragm], implants, injectable or oral contraceptives [must have been using for at least the last 3 months], some intrauterine contraceptive devices, tubal ligation, or in an established relationship with a vasectomized partner) during the entire duration of the study
* Be willing to maintain stable dietary habits and physical activity levels throughout the trial period;
* Be able to communicate well with the Investigator, to understand and comply with the requirements of the study and be judged suitable for the study in the opinion of the Investigator.

Within 3 months following to the exit of the study for failure to comply with one or more of the inclusion criteria listed above, a re-screening could be performed.

Exclusion Criteria:

* Uncontrolled hyperglycemia assessed by HbA1c ≥ 6.5%;
* Suffering from a metabolic disorder such as diabetes mellitus that requires lifesyle and dietary recommendations or a medication according to the recommendations, uncontrolled thyroidal trouble (Confirmed by clinical significant abnormal TSG/T4 and/or stabled medication for >3 months) or other metabolic disorder;
* Suffering from a severe chronic disease (e.g., cancer, HIV, renal failure, hepatic or biliary disorders ongoing, chronic inflammatory digestive disease, inflammatory bowel disease, irritable bowel syndrome, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g., celiac disease);
* With a history of retinopathy, microalbuminuria, ischemic cardiovascular event during the previous 6 months;
* Consumption of more than 30 g of dietary fibre per day, as measured by the Block Fibre Screener
* Prior diagnosis of Type I diabetes mellitus (i.e., a clinical diagnosis made before the screening visit of this study);
* Alcohol consumption (>21 units per week);
* Smoking more than 10 cigarettes per day;
* Previous bariatric surgery;
* Any surgery in the 3 months before the study or planned for 6 months after enrolling;
* Pregnancy or pregnancy planned in the 6 months after enrolling or lactating women;
* Consumption of dietary supplements (omega-3 fatty acids, probiotics, prebiotics, plant stanols/sterols) in the 4-weeks before the study;
* Presence or history of significant and diagnosed gastrointestinal diseases that, in the opinion of the investigator, could be associated with disturbed gastrointestinal absorption (e.g., resections, diverticula, active and diagnostically confirmed irritable bowel syndrome, malabsorption syndrome);
* Present or recent (within 3-months of screening) use of any other medication which, in the opinion of the investigator, could interfere with the outcome of the study, including but not limited to antithrombotic agents, anti-inflammatory agents and chronic NSAID use (except low-dose prophylactic, proton pump inhibitors (PPIs), antihistamines, if ongoing (3-months) and on a stable dose throughout study period);
* Steroids (over the counter (OTC) NSAIDS, topical steroids and inhalers are allowed)
* Current or planned participation in a weight-loss regimen (including intermediate fasting), including extreme dietary practices or exercise;
* Anorexia nervosa, bulimia or significant eating disorders according to the investigators;
* Having lost >5% of their body weight within 3-months prior to screening;
* Lactose intolerance or milk protein allergy;
* Gluten intolerance;
* Current treatment with medications influencing the parameters of interest (glucose-lowering drugs such as metformin, DPP4 inhibitors, GLP-1 receptor agonists, acarbose, sulfonylureas, glinides, thiazolidinediones, sodium-glucose cotransporter -2 inhibitors, insulin, lactulose, glucocorticoids, immunosuppressive agents, , orlistat, cholestyramine or ezetimibe);
* Antibiotic use in the 3 months before the study;
* Participant has a known allergy to inactive or active ingredients in the study products;
* Participation in other clinical research trials within 90 days prior to randomization;
* Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity by Matsuda Index | From baseline to day 120
  Absolute change from baseline to day 120 in treatment group as compared to placebo in insulin sensitivity as determined by Matsuda.

SECONDARY OUTCOMES:
Insulin sensitivity by homeostasis model assessment-estimated (HOMA) insuline sensitivity | From baseline to day 120
  change in treatment group as compared to placebo by measuring fasting glucose and insulin values
fasting blood glucose | From baseline to day 120
  change in treatment group as compared to placebo
3-hour blood glucose incremental Area Under the Curve (AUC) as measured by Oral Glucose Tolerance Test (OGTT) | From baseline to day 120
  change in treatment group as compared to placebo
Peak Plasma Concentration (Cmax) of blood glucose as measured by OGTT | From baseline to day 120
  change in treatment group as compared to placebo
3-hour blood insulin incremental Area Under the Curve (AUC) as measured by OGTT | From baseline to day 120
  change in treatment group as compared to placebo
Peak Plasma Concentration (Cmax) of blood insulin as measured by OGTT | From baseline to day 120
  change in treatment group as compared to placebo
Glycosylated hemoglobin (HbA1c) | From baseline to day 120
  change in treatment group as compared to placebo
Postprandial triglyceride (TG) response as incremental Area Under the Curve (AUC) as measured by OGTT | From baseline to day 120
  change in treatment group as compared to placebo
Peak Plasma Concentration (Cmax) of blood TG as measured by OGTT | From baseline to day 120
  change in treatment group as compared to placebo
Blood lipid profile by total cholesterol, TG, low density lipoprotein, high density lipoprotein, non-esterified fatty acids | From baseline to day 120
  change in treatment group as compared to placebo
Liver enzymes (ALT, AST, GGT, bilirubin, alkaline phosphatase) | From baseline to day 120
  change in treatment group as compared to placebo
Anthropometry by Height (m) and body weight (kg) combined into BMI (kg/m2) | From baseline to day 120
  change in treatment group as compared to placebo
Circumference (cm) of waist, hip and neck and waist, hip and height measurement will be combined into Waist-to-Hip ratio (W:H) and Waist-to-Height ratio (WHtR) | From baseline to day 120
  change in treatment group as compared to placebo
Body composition by measurement of body fat mass by DEXA measurement | From baseline to day 120
  change in treatment group as compared to placebo
Body composition by measurement of lean mass by DEXA measurement | From baseline to day 120
  change in treatment group as compared to placebo
Body composition by measurement of trunk fat mass by DEXA measurement | From baseline to day 120
  change in treatment group as compared to placebo
Vital signs: heart rate | From baseline to day 120
  evaluation of heart rate
Vital signs: blood pressure | From baseline to day 120
  evaluation of Systolic blood pressure (SBP) (mmHg) and diastolic blood pressure (DBP) (mmHg)
Vital signs: body temperature | From baseline to day 120
  evaluation of body temperature
Vital signs: respiratory rate | From baseline to day 120
  evaluation of respiratory rate
Adverse events | From baseline to day 120
  evaluation of occurrence of the nature, frequency, severity and relatedness of adverse events as well as clinically significant laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Peter Suenaert, MD, PhD, Study Director — R&D and Clinical Development
Locations (2):
- Clinical Research Center (CRC) Kiel GmbH, Kiel, Germany
- Atlantia Food Clinical Trials, Cork, Ireland

REFERENCES:
- [Background] Depommier C, Everard A, Druart C, Plovier H, Van Hul M, Vieira-Silva S, Falony G, Raes J, Maiter D, Delzenne NM, de Barsy M, Loumaye A, Hermans MP, Thissen JP, de Vos WM, Cani PD. Supplementation with Akkermansia muciniphila in overweight and obese human volunteers: a proof-of-concept exploratory study. Nat Med. 2019 Jul;25(7):1096-1103. doi: 10.1038/s41591-019-0495-2. Epub 2019 Jul 1. PMID 31263284